CLINICAL TRIAL: NCT01773785
Title: Phase II Study of SPI-1620 in Combination With Docetaxel as a Second-Line Treatment for Patients With Advanced Biliary Cancer
Brief Title: Phase II Study of SPI-1620 in Combination With Docetaxel as a Second-Line to Treat Biliary Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study completed the first phase and did not meet efficacy end point to enter into the randomized phase.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-1620-12-202
Record Dates: First submitted 2013-01-14; First posted 2013-01-23 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Biliary Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — sovateltide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPI-1620 & Docetaxel (Experimental): Patients will receive 11 μg/m2 of SPI-1620 intravenously over one minute. Ten minutes after (±2 min) SPI-1620 administration, patients will receive docetaxel 75 mg/m2 intravenous. This regimen will be repeated every 3-weeks cycles until progression or intolerable toxicity.
  Interventions: Drug: SPI-1620; Drug: Docetaxel

INTERVENTIONS:
Drug: SPI-1620 — SPI-1620 11 μg/m2 will be given intravenously over 1 minute.
Drug: Docetaxel — Docetaxel 75 mg/m2 infusion will be administered per standard of care 10 (±2) minutes after SPI-1620.

SUMMARY:
The primary purpose of this study is to determine the effectiveness of SPI-1620 in combination with docetaxel in patients with advanced biliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed biliary tract or gallbladder cancer that have relapsed or are refractory after one prior gemcitabine-based chemotherapy regimen for advanced biliary cancer
* Evaluable disease
* ECOG PS ≤ 2
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Treatment with more than one prior chemotherapy regimen
* Known, uncontrolled CNS metastases
* Baseline peripheral neuropathy ≥ grade 2.
* Significant circulatory disorders in the past 6 months
* Concomitant use of phosphodiesterase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 18 months

SECONDARY OUTCOMES:
Overall response rate | 18 months
Overall survival | 18 months
Duration of Response | 12 months
Safety of SPI-1620 when administered in combination with docetaxel | 12 months
  Periodic physical examinations with vital sign monitoring, safety laboratories and monitoring of adverse events will be performed

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Miami Hospitals & Clinics/ Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington